CLINICAL TRIAL: NCT06824272
Title: The Effect of a Hybrid Support Program Based on the Hypnofertility and Health Improvement Model on Infertile Women's Fertility Readiness, Self-Efficacy, Lifestyle, and Pregnancy Outcomes
Brief Title: Online and Mobile Support Program and Fertility
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, ESRA ARBAG, nurse, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DEU-HF-FY-OI
Record Dates: First submitted 2025-01-20; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Infertility; Stress
Keywords: Hypnofertility; Fertility Preparedness; Self-efficacy; Lifestyle; Pregnancy Outcome; Mobile Application; Online Education; infertility; pender
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Our study includes an experimental group and a control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Before the first lesson of the online fertility preparation class, the Informed Voluntary Consent Form, the Introductory Information Form, the Fertility Readiness Scale for Women Receiving Fertility Support, the Infertility Self-Efficacy Scale-Short Form (İÖYÖ-KF) and the Healthy Lifestyle Behaviors Scale for Enhancing Fertility will be administered to the women. After the online fertility preparation class is applied synchronously in groups for four weeks, the Fertility Readiness Scale, the Infertility Self-Efficacy Scale-Short Form (İÖYÖ-KF) and the Healthy Lifestyle Behaviors Scale for Enhancing Fertility will be administered to the women again in the last session. After the online fertility preparation classes, the women will start IVF treatment. At this stage, the Fertility Readiness Scale for Women Receiving Fertility Support, the Infertility Self-Efficacy Scale-Short Form and the Healthy Lifestyle Behaviors Scale for Improving Fertility will be administered to the women again.
  Interventions: Other: MOBIL AND ONLINE EDUCATION
- Control (No Intervention): The control group will not receive any training. They will undergo routine IVF treatment. On the 2nd or 3rd day of the cycle, which is the first day of treatment, the Informed Consent Form, the Informational Brochure, the Fertility Readiness Scale for Women Receiving Fertility Support, the Infertility Self-Efficacy Scale - Short Form (ISF-SF), and the Healthy Lifestyle Behaviors Scale for Improving Fertility will be administered. One to two days before the pregnancy test, the Fertility Readiness Scale for Women Receiving Fertility Support, the Infertility Self-Efficacy Scale - Short Form (ISF-SF), and the Healthy Lifestyle Behaviors Scale for Improving Fertility will be administered again to the women. The results of the pregnancy test will be recorded, and the steps to be taken for the control group will be concluded.

INTERVENTIONS:
Other: MOBIL AND ONLINE EDUCATION — The intervention group attended synchronous online sessions twice weekly (2 hours) for four weeks before IVF, with the mobile app available from the first session. During IVF cycles, the app provided scheduled educational content, reminders, creation of lifestyle maps, feedback,counseling scheduling, and daily motivational messages based on hypnofertility principles to enhance support.
  Arms: Intervention

SUMMARY:
Our study is designed as a randomized controlled experimental study with a pre-test and post-test control group to determine the effects of online fertility preparation classes and fertility mobile application support, based on the Philosophy of Hypnofertility and Pender's Health Promotion Model, on infertile women's fertility readiness, fertility self-efficacy, lifestyle, and pregnancy outcomes.

DETAILED DESCRIPTION:
The research will be conducted with women who apply for infertility treatment at institutions providing such services in İzmir (İzmir Dokuz Eylul University Hospital, İzmir Ege Maternity and Women's Diseases Training and Research Hospital, İzmir Medical Park Hospital) and who agree to participate in the study and meet the sampling criteria. It is planned that the training, based on the philosophy of Hypnofertility and Pender's Health Promotion Model, will be conducted in the form of synchronous remote education through online fertility preparation classes created by the researchers. Additionally, a Fertility mobile application will be developed. In our study, training will be provided on healthy lifestyle changes for fertility, including physical activity, sleep, nutrition, and stress management. The investigators have based the content of our training on Pender's Health Promotion Model. Thus, the investigators believe that our training will help women become aware of the relationship between their health status and health behaviors, and by empowering them to change behaviors that negatively affect their fertility, the investigators will enhance health-promoting behaviors. During our training sessions, the investigators will collect data related to women's previous behaviors, personal factors (biological, psychological, and sociocultural), self-efficacy, perceived benefits, and barriers. Based on the collected data, the investigators will create a health promotion plan that takes into account the individual's past experiences, personal factors, perceived barriers, self-efficacy issues, emotional challenges, and perceived benefits of action. In the implementation phase, the investigators will ensure that individuals incorporate health-promoting behaviors into their lives and routines. In this way, the investigatorsbelieve that the training the investigators provide will contribute to making these behaviors a part of individuals' lifestyles. the investigators will use Pender's health promotion model in our training sessions as follows. For example, let's consider the topic of examining the impact of our lifestyle habits on fertility and questioning behaviors that promote fertility. The investigators will investigate the physical activity status of individuals, learning about the perceived benefits and barriers they associate with engaging in moderate physical activity, which is a healthy lifestyle behavior that enhances fertility. Based on this information, the investigators will create a program that supports individuals in incorporating moderate physical activity into their daily routines, and the investigators will even enhance this with a mobile application. Our goal here is to reduce the perceived barriers to health-promoting behaviors and increase the perceived benefits, enabling individuals to integrate health-enhancing behaviors into their lives and routines during the implementation phase. In this way, the investigators believe that by influencing the urgent needs and choices under the behavioral outcomes of Pender's model, the training the investigators provide will contribute to making these behaviors a part of individuals' lifestyles.A class will be opened when the number of women is at least 3 and at most 7. The online fertility preparation classes are aimed to be conducted synchronously during the first four weeks before the women begin IVF treatment. The synchronous part of the program is planned to be four weeks long, with two days a week and two-hour sessions (eight sessions in total). A software company will be engaged to transfer the presentations, written materials, relaxation audio recordings, and fertility massage videos into a mobile application using Android programming for the online fertility preparation classes.The organization, compliance, presentation, interaction, and navigation elements will be taken into account in the creation of the mobile application. The mobile application is planned to be designed in a simple and user-friendly organizational structure to appeal to all women as much as possible. The usability of the mobile application created on the Android platform will be tested on 5 couples who are not included in the research sample to ensure control. Couples in the intervention group will be able to download the mobile application from Playstore and App Store to their phones and start using it from the first meeting. Usernames and passwords will be created for the women in this group for their login processes. While women can use the mobile application at any time they wish, there are educational videos and audio recordings they need to follow at specific times during their treatment cycles (the first folliculometry day, the second folliculometry day, OPU day, and embryo transfer day). After women register their treatment start times in the application, they will be reminded of the educational videos they need to follow through notifications sent by the application. This application will also include a management panel where the researcher can track the women's lifestyle maps. The researcher will be able to log into this panel with a username and password to provide feedback to the women regarding their lifestyle maps (physical activity, sleep, nutrition, and stress). Additionally, the application will feature a panel where they can ask questions to the researcher and a section where they can specify the day and time they would like to receive individual counseling if they wish to do so synchronously. The mobile application will automatically send positive messages that enhance motivation, aligned with the language of hypnofertility, to women every day.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with primary infertility,

  * Having been diagnosed with female, male factor and unexplained infertility,
  * Cycles where fresh embryos will be applied
  * Having In Vitro Fertilization (IVF) treatment,
  * Knowing how to read and write Turkish,
  * Being able to use a computer, internet and mobile phone
  * Having a smart phone,
  * Being able to use a smart phone,
  * Having internet access,
  * Agreeing to participate in the study

Exclusion Criteria:

* Cycles to be performed with frozen embryos

  * Having any psychiatric disorder,
  * Attending less than 80% of the trainings (not attending more than 2 classes) in this case women will be excluded from the study and in order to reach a sufficient sample, institutions will be visited again and cases that meet the sample criteria will be found. Re-randomization will be done among women who meet the criteria
  * Having any chronic disease for which they are receiving treatment.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — women
Enrollment: 128 (Estimated)
Dates: Start 2025-03-30 (Estimated); Primary Completion 2025-08-12 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
pregnancy outcome | 1 mounth
  The occurrence of clinical pregnancy after treatment will be evaluated.

SECONDARY OUTCOMES:
Fertility Readiness, Self-efficacy, Lifestyle | 6 mounth
  Fertility Readiness Scale for Women Receiving Fertility Support; A high score indicates strong fertility readiness. The minimum score that can be obtained from the scale is 23, while the maximum score is 115.

OTHER OUTCOMES:
Fertility Self Eficacy | 6 mounth
  The Infertility Self-Efficacy Scale - Short Form (ISSS-SF) scores range from 8 to 32. As the score increases, the perception of self-efficacy is considered to be higher. All statements in the scale are positively worded, and there is no cutoff point for the scale.
Healthy Lifestyle Behaviors | 6 mounth
  The 46-item Scale of Healthy Lifestyle Behaviors in Fertility Development is scored on a 5-point Likert scale, with a minimum score of 46 and a maximum score of 230. An increase in the scale score indicates a higher intensity of healthy lifestyle behaviors among individuals.

CONTACTS AND LOCATIONS:
Overall Officials: DEU, Study Director — DEU

IPD SHARING:
Plan to Share IPD: No